CLINICAL TRIAL: NCT00781976
Title: A Randomised, DB, PC Study to Determine the PK, Safety and Tolerability Profile and Antiviral Activity of Multiple Oral Doses of AZD7295 in Otherwise Healthy Male and Female Hepatitis C Carriers With Compensated Liver Disease
Brief Title: Antiviral Activity of AZD7295 in HCV Carriers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrow Therapeutics (Industry)
Responsible Party: Liz Clark, Arrow Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCV689-102
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: AZD7295

INTERVENTIONS:
Drug: AZD7295 — 700mg per day maximum
  Arms: 2
Drug: Placebo — matched placebo
  Arms: 1

SUMMARY:
PK, safety study of AZD7295 in HCV carriers

ELIGIBILITY:
Inclusion Criteria:

* HCV carrier

Exclusion Criteria:

* concurrent medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Plasma AZD7295 concentrations and pharmacokinetics | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Ed Gane, Principal Investigator — Auckland Clinical Services
Locations (1):
- Prof Ed Gane, Auckland, New Zealand